CLINICAL TRIAL: NCT01019681
Title: Umbilical Cord Blood Stem Cell Injection for Critical Limb Ischemia
Brief Title: Efficacy and Safety of Umbilical Cord Blood Injection for Critical Limb Ischemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Only patient enrolled on study died -the cause of death not study related
Sponsor: Richard Burt, MD (Other)
Responsible Party: Sponsor-Investigator, Richard Burt, MD, MD, Northwestern University
Organization: Northwestern University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PVD.Cord.Blood.2008
Record Dates: First submitted 2009-11-19; First posted 2009-11-25 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Critical Limb Ischemia
Keywords: Cord blood injection in peripheral vascular disease
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UBC injection into one leg of PVD pt (Experimental): 25 participants with severe peripheral vascular disease in leg(s) and they do not qualify for surgical treatment.
  Interventions: Biological: Cord blood stem cell injection

INTERVENTIONS:
Biological: Cord blood stem cell injection — The cord blood stem cells will be simply injected intramuscularly in the leg. 30 minutes prior to stem cell injection the patients will receive Vancomycin 1 gram IVPB x1 as a prophylactic measure. Patients will also receive Ativan 0.5 to 1 mg PO x 1 and Dilaudid 0.5 to 1 mg IV x1 to alleviate the discomfort of the procedure.
  Cells will be injected by means of a 22 gauge sterile spinal needle after topical anesthesia of the injection site. The concentration will be at least 2 x 107 total nucleated cells per ml in phosphate buffered saline (PBS) with 5% human serum albumin (Baxter, Deerfield Illinois).
  Other Names: HSCT

SUMMARY:
The purpose of this study is to determine whether treatment with umbilical cord blood stem cells will improve blood flow to the most severely affected leg of a participant with medically refractory and non-surgical peripheral vascular disease of the lower extremity.

DETAILED DESCRIPTION:
Umbilical cord blood is a safe alternative source of stem cells used for decades in hematopoietic stem cell transplants for malignancies. There is also a reported decreased incidence of acute GVHD compared to matched unrelated donor transplants.A cord blood registry will be searched for suitable units with compatibility in the ABO and HLA systems. The minimum total nucleated cell dose required which would be 1.0 x 107/kg, and one unit of cells will be procured to meet this requirement. Although it is likely that the transplanted cord blood cells will be rejected over time, we hypothesize that while they remain in the host's tissue these cells will be producing and releasing cytokines, growth factors and other humoral factors that might promote vasculogenesis by stimulating endogenous stem cells and endothelial cells. Since there is no need to collect the patient's own stem cells, the patient's cardiovascular system will not be subjected to any stress due to the leukapheresis procedure itself. No injections of exogenous growth factors, which have been associated with thrombosis, would be required to mobilize the patient's own stem cells. The procedure could conceivably even be performed in its entirety on an outpatient basis.

A total of 25 patients will be enrolled in the study. Patients will be followed for 24 months after the procedure with evaluation visits one day after the transplant and then at one month, six, twelve and twenty four months post-treatment. The visit one day after the transplant will involve a history and physical with a leg exam, a CBC and a chemistry panel to evaluate for possible infection, or other adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Atherosclerotic ischemic peripheral vascular disease or Thromboangiitis Obliterans with Critical Limb Ischemia (Fontaine stages III and IV)
* Participant must match either a or b

  1. Ankle brachial index (ABI) ≤ 0.7
  2. Doppler waveforms at posterior tibial artery and dorsalis pedis artery are monophasic with toe pressure < 30 mmHg.
* A non-surgical candidate for revascularization e.g. prior vascular reconstruction, inability to locate a suitable vein for grafting, diffuse multi- segment disease, or extensive infra-popliteal disease not amenable to a vascular graft.
* Age > 18 years old.
* The non-index leg may be treated only in the event and it full fills the same eligibility criteria and exclusion criteria used in this protocol for the treatment leg.
* Patients must be on maximal tolerated medical therapy for PVD including A) Cessation of smoking B) Referral to endocrinologist for control of HgA1c to < 7.0 mg/dl, control of hyperlipidemia with statins or other anti-hyperlipidemic drugs as indicated, control of hypertension as indicated C) Antiplatelet therapy with aspirin and / or cilostazol (unless medically contraindicated, e.g. bleeding or allergy)

Exclusion Criteria:

* Popliteal vascular entrapment syndrome
* Lower extremity infection or infected ulcer
* Hypercoagulable state
* HIV positive
* HBsAg positive
* Uncontrolled arrhythmia, that is, persistence of an arrhythmia despite medical therapy
* Unstable angina
* Thrombocytopenia < 50,000/ul
* Leukemia or myelodysplasia
* Allergy to E coli or its products
* Patients with metal in their bodies cannot undergo MRIs (MRA). Therefore, patients with, cochlear implants, or aneurysm clips are not eligible. Coronary artery stents are not a contraindication. Patients with pacemakers are still candidates provided they have normal creatinine (< 1.1 mg/dl) and can receive contrast dye (no allergy) for angiogram instead of MRA. MRI/MRA does not need to be repeated if a prior MRA or Angiogram Demonstrates inoperable disease.
* Patients who are pregnant
* Poorly controlled diabetes will not be a cause for exclusion but patient must see endocrinologist for better control
* Current malignancy, except squamous cell or basal cell skin cancers thought to be easily controlled.
* AST, ALT, or bilirubin more than twice the upper limit of normal.
* WBC < 2.5 / ul.
* Any patient who is actively bleeding, including blood on urine dipstick or fecal occult blood.
* Patient is on chemotherapy or other immuno-suppressive medications such as steroids, cellcept, cyclosporine, cytoxan, azathioprine, rituxan, humira or remicade.
* Donor is HLA homozygous and shares that HLA haplotype with the recipient (a different donor will have to be found)
* Patients diagnosed with Thromboangiitis Obliterans (Buerger's Disease) who are smokers and are unwilling or unable to quit smoking
* A) Patients with a myocardial infarction within the last 30 days or left ventricular ejection fraction < 35% B) Patients with a history of malignancy in the last 5 years (other than basal cell carcinoma or carcinoma in situ) C) Patients with a CVA within the last 6 months D) Patients with a HbA1c level > 7.0%

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Ankle brachial index (ABI), a 15% increase will be considered improvement | Pre-transplant, 1, 6, 12 and 24 months after
Healing of ischemic ulcers | Pre-transplant, 1, 6, 12 and 24 months after
Decreased pain level as reported by the patient | Pre-transplant, 1, 6, 12 and 24 months after

SECONDARY OUTCOMES:
SF-36 quality of life (QOL) | Pre-transplant, 1, 6 , 12, and 24 months after HSC transplant
Walking Impairment Questionnaire | Pre-transplant, 1, 6 , 12, and 24 months after HSC transplant
Increase in pain free ambulation time on treadmill by more than 25% | Pre-transplant, 1, 6 , 12, and 24 months after HSC transplant
Increase in four meter walk or six minute walk by more than 25% | Pre-transplant, 1, 6 , 12, and 24 months after HSC transplant

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University and Northwestern Memorial Hospital
Locations (1):
- Northwestern University, Chicago, Illinois, United States